CLINICAL TRIAL: NCT06199752
Title: Synergistic Immunomodulatory Effect of Synbiotics Pre and Postoperative Resection of Pancreatic Ductal Adenocarcinoma
Acronym: PDAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Maher Sara, Dr, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Synbiotics in cancer
Record Dates: First submitted 2023-11-29; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Active Comparator): Placebo consisted of identical capsules of powdered glucose polymer
  Interventions: Dietary Supplement: probiotic agent 25 Billion CFU (Nowfoods, USA) , ). Inulin capsules 1000mg Herbamama USA
- Synbiotics group (Placebo Comparator): probiotic agent 25 Billion CFU (Nowfoods, USA), + Inulin capsules 1000mg two capsules once daily. Herbamama USA
  Interventions: Dietary Supplement: probiotic agent 25 Billion CFU (Nowfoods, USA) , ). Inulin capsules 1000mg Herbamama USA
- Probiotics group (Placebo Comparator): probiotic agent 25 Billion CFU (Nowfoods, USA)
  Interventions: Dietary Supplement: probiotic agent 25 Billion CFU (Nowfoods, USA) , ). Inulin capsules 1000mg Herbamama USA

INTERVENTIONS:
Dietary Supplement: probiotic agent 25 Billion CFU (Nowfoods, USA) , ). Inulin capsules 1000mg Herbamama USA — probiotic agent 25 Billion CFU (Nowfoods, USA), composed of ten strains of bacteria (Lactobacillus acidophilus, Bifidobacterium lactis, Lactobacillus plantaLactobacillus paracasei, Bifidobacterium breve, Streotococcus thermophiles, Lactobacillus salivarius, and Bifidobacterium longum),

SUMMARY:
The goal of this interventional study was to evaluate the synergistic effect of symbiotics (a combination of probiotics and prebiotics) compared to probiotics alone in terms of their impact on anti-tumor immunomodulation in patients with pancreatic ductal adenocarcinoma (PDAC). The study also aimed to assess the effects of these interventions on postoperative complications and outcomes. In the study, a probiotic agent (Nowfoods, USA), containing ten strains of bacteria with a total dosage of 25 billion colony-forming units (CFU) was administered. This probiotic regimen involved taking two capsules once daily, starting two weeks before the surgery and continuing for one month after the surgery. For the synbiotic group, in addition to the probiotic agent, two capsules per day of inulin supplement (HERBAMAMA, USA) were also taken.

The study included three groups: the synbiotics group, the probiotics group, and the placebo group. The researchers compared the pathological status of immune cell infiltration (specifically CD8 cells) and interferon-gamma expression, as well as the levels of interleukins 10, 6, and 10 in the participants' serum. Four blood samples were collected from each participant: one taken 14 days before the surgery, one on the surgery date, one two weeks after the surgery, and one 30 days after the surgery.

The main research question addressed by the study was whether there was a significant difference in the immunomodulatory effect and postoperative complications between the synbiotics group and the probiotics group. The placebo group likely served as a control to compare the effects of the interventions against no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary PDAC with complete pathological and follow-up data
* Patients without long-distance metastasis
* Patients without chronic diseases
* Patients without any treatments before the surgery.

Exclusion Criteria:

* Patients who suffered from other tumors or other chronic diseases or accidentally died
* Lack of pathological and follow-up data.
* Patients with long-distance metastasis before the surgery.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-12-12 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Immunohistochemistry testing for immune cells infiltration and interferon-gamma expression | IHC testing for formalin fixed paraffin embedded block for all subjects 10 months from the beginning of the study, as we collected the all samples
  Change in the percentage of infiltrating CD8T cells in the tumor tissue as well as the interferon-gamma in synbiotics group
Inflammatory cytokines level | 10 months after collection of all blood samples from included subjects
  A change in the inflammatory cytokines levels (IL 10, IL6, and IL 1 β) in synbiotics-treated group with a significant difference rather the placebo and probiotics only treated groups
Post-operative -non-infectious complications- improvement | 1-4 weeks post operative
  Testing the percentage of subjects having Anastomotic Leakage, Diarrhea, Abdominal distension
Post-operative -infectious complications improvement | 1-4 weeks post operative
  Testing the percentage of subjects having Bacteremia, Wound infection, Pneumonia, Urinary tract infection
Post-operative improvement days | first day post operative till 20 days
  Number of days for first stool, stay in the hospital and return to usual activity
Statistical analysis of the results | 11 months from the beginning of the study
  To assess the significance of changes in the percentage of CD8 cells in the tissue in all subjected groups as well as the expression of Interferon-gamma protein. Also, the concentration of circulating cytokines including IL B, IL6, and IL 10.
  Data were analyzed using statistical software package (IBM-SPSS) version 23 software. Kolmogorov-Smirnov test showed that the raw data were normally distributed. One ANOVA was applied to study the effect of treatment on the studied parameters. Two-way ANOVA was applied to study the effect of time and treatment on the studied parameters. The least significant difference (LSD) test was used to illustrate the statistical differences among the experimental groups. Duncan's test was used to illustrate the homogeneity among the different intervals. Data is displayed as mean ± standard error of the mean.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Maher, Principal Investigator — Theodor Bilharz Research Institute
Locations (1):
- Sara Maher, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sobocki BK, Kazmierczak-Siedlecka K, Folwarski M, Hawrylkowicz V, Makarewicz W, Stachowska E. Pancreatic Cancer and Gut Microbiome-Related Aspects: A Comprehensive Review and Dietary Recommendations. Nutrients. 2021 Dec 10;13(12):4425. doi: 10.3390/nu13124425. PMID 34959977
- [Derived] Maher S, Elmeligy HA, Aboushousha T, Helal NS, Ossama Y, Rady M, Hassan AMA, Kamel M. Synergistic immunomodulatory effect of synbiotics pre- and postoperative resection of pancreatic ductal adenocarcinoma: a randomized controlled study. Cancer Immunol Immunother. 2024 Apr 25;73(6):109. doi: 10.1007/s00262-024-03686-6. PMID 38662232

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT06199752/Prot_SAP_000.pdf